CLINICAL TRIAL: NCT04760860
Title: a Randomized, Double Blind, Placebo Controlled Clinical Trial Exploring the Target Engagement and Tolerability of Terazosin Hydrochloride in Patients With Dementia With Lewy Bodies
Brief Title: Terazosin for Dementia With Lewy Bodies
Acronym: TZ-DLB
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qiang Zhang (Other)
Responsible Party: Sponsor-Investigator, Qiang Zhang, Associate of Neurology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202101470
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Dementia With Lewy Bodies
MeSH Terms: conditions — Lewy Body Disease | interventions — Terazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo Control Arm (Placebo Comparator): Participants in this arm will receive placebo during the trial for 15 weeks, the placebo will follow the same schedule as the Terazosin group; the placebo capsules will have the same appearance as the Terazosin capsules.
  Interventions: Other: Placebo
- Terazosin Arm (Experimental): Participants in this arm will receive Terazosin during the trial for 15 weeks. Participants will start at 1mg daily for the first 6 week, then the dosage will be increased to 5mg daily over 3 weeks, and continued for the last 6 weeks.
  Interventions: Drug: Terazosin Hydrochloride

INTERVENTIONS:
Drug: Terazosin Hydrochloride — In this double blind, randomized, placebo controlled phase I clinical trial, subjects randomized into the Terazosin group will receive Terazosin hydrochloride treatment for 15 weeks. Participants will start at 1mg daily for the first 6 week, then the dosage will be increased to 5mg daily over 3 weeks, and continued for the last 6 weeks.
  Other Names: Terazosin, Hytrin
  Arms: Terazosin Arm
Other: Placebo — In this double blind, randomized, placebo controlled phase I clinical trial, subjects randomized into the control group will receive placebo for 15 weeks.
  Arms: Placebo Control Arm

SUMMARY:
The TZ-DLB trial will be a 3:2 (active:placebo) randomized, double-blind, placebo-controlled Pilot trial to evaluate the tolerability of terazosin for the treatment of dementia with Lewy bodies.

DETAILED DESCRIPTION:
This will be a single center, randomized, double-blind, placebo-controlled, pilot study to assess the tolerability of terazosin (TZ) at 1 and 5 milligrams (MG) daily for patients with DLB. The primary goal of this study is to assess the tolerability of TZ in patients with DLB. This is a pilot study and is not powered to assess efficacy of this medication. Our hope is that this study will guide future studies of this (and similar) medications for the disease modification of DLB. This study is also aimed to learn more about how patients with produce and use energy and if TZ can help to reverse energy deficits that appear in DLB.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with the diagnosis of dementia with Lewy Bodies per 2017 DLB Consortium criteria.
* Baseline MOCA 18 or above. On stable AChEI and/or memantine treatment regimen for ≥4 weeks prior to baseline.

Exclusion Criteria:

* Subjects unwilling or unable to give informed consent
* No confounding acute or unstable medical, psychiatric, orthopedic condition. Subjects who have hypertension, diabetes mellitus, depression, or other common age-related illness will be included if their disease under control with stable treatment regimen for at least 30 days.
* Orthostatic hypotension defined as symptomatic decrease in BP > 20mmHg systolic or > 10mmHg diastolic on supine to sitting or standing, or a sitting blood pressure of ≤90/60.
* Clinically significant traumatic brain injury or post-traumatic stress disorder
* Presence of other known medical comorbidities that in the investigator's opinion would compromise participation in the study
* Psychiatric comorbidities including major depression, bipolar affective disorder, or other mental health disorders that are sufficiently severe to increase adverse event risk or impact neurology assessment in the opinion of the responsible site principal investigator. Subjects with clinically significant depression as determined by a Beck Depression Inventory score greater than 21 at the screening visit. Current suicidal ideation within one year prior to the baseline visit as evidenced by answering "yes" to Questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale (C-SSRS) If the participant has a Beck Anxiety Score greater than 22 at the initial screening visit.
* Use of investigational drugs within 30 days before screening
* Subjects have to be on a stable regimen of central nervous system acting medications (benzodiazepines, antidepressants, hypnotics) for 30 days prior to the baseline visit
* Use of doxazosin, alfuzosin, prazosin, or tamsulosin
* For female participant, pregnancy, or plans for child-bearing during study period
* Participant is restricted from traveling to and from the study site

Ages: 0 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of intervention-related adverse events between treatment arms | 15 weeks
  All patient-reported adverse events will be compared.
Frequency of drop-out/discontinuation of study intervention for any reason | 15 weeks
  The number of participants in each group who drop out of the study for any reason will be compared.
Brain [ATP] as measured by 31P-Magnetic Resonance Spectroscopy | at baseline, 6 weeks and 15 weeks
  Brain [ATP] as measured by 31P-Magnetic Resonance Spectroscopy

SECONDARY OUTCOMES:
To assess the mean change in systolic and diastolic blood pressures | at baseline, 6 weeks and 15 weeks
  Blood pressure will be evaluated at baseline, 2 weeks, 6 weeks and 12 weeks
Unified Parkinson Disease Rating Scale (UPDRS) part III Motor examination | at baseline, 6 weeks and 15 weeks
  Unified Parkinson Disease Rating Scale (UPDRS) part III will be evaluated at baseline, 2 weeks, 6 weeks and 12 weeks
Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) | at baseline, 6 weeks and 15 weeks
  Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) will be evaluated at baseline and 12 weeks
Montreal Cognitive Assessment | at baseline, 6 weeks and 15 weeks
  Montreal Cognitive Assessment
The Clinician Interview-Based Impression of Change, plus carer interview (CIBIC-Plus) | at baseline, 6 weeks and 15 weeks
  CIBIC-Plus will be evaluated at baseline and at 12 weeks
Neuropsychiatric inventory | at baseline, 6 weeks and 15 weeks
  NPI will be evaluated at baseline and at 12 weeks
Fluorodeoxyglucose (FDG)-positron emission tomography (PET) | at baseline, 6 weeks and 15 weeks
  A surrogate for glucose metabolism in the brain
Serum ATP levels | at baseline, 6 weeks and 15 weeks
  Serum ATP level changes will be compared between the TZ and the placebo arms
Serum TeraZosin levels | at baseline, 6 weeks and 15 weeks
  Serum Terazosin levels will be analyzed and a correlation between ATP levels and TZ levels will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Nandakumar Narayanan, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request with justification for request from qualified researchers, anonymized data will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year after completion of this study
Access Criteria: Qualified researchers may contact the PI of this study with reasonable requests for data to be shared. Inquiries must include what hypothesis the researcher intends to test using the shared data.

REFERENCES:
- [Background] Cai R, Zhang Y, Simmering JE, Schultz JL, Li Y, Fernandez-Carasa I, Consiglio A, Raya A, Polgreen PM, Narayanan NS, Yuan Y, Chen Z, Su W, Han Y, Zhao C, Gao L, Ji X, Welsh MJ, Liu L. Enhancing glycolysis attenuates Parkinson's disease progression in models and clinical databases. J Clin Invest. 2019 Oct 1;129(10):4539-4549. doi: 10.1172/JCI129987. PMID 31524631
- [Background] Simmering JE, Welsh MJ, Liu L, Narayanan NS, Pottegard A. Association of Glycolysis-Enhancing alpha-1 Blockers With Risk of Developing Parkinson Disease. JAMA Neurol. 2021 Apr 1;78(4):407-413. doi: 10.1001/jamaneurol.2020.5157. PMID 33523098